CLINICAL TRIAL: NCT05713487
Title: Preventive Treatment of Groin Pain Syndrome in élite Young Football Player: a Pilot Study
Brief Title: Preventive Treatment of Groin Pain in Football
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Luca Puce, principal investigator, Universita degli Studi di Genova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GP-DINOGMI-23
Record Dates: First submitted 2023-01-24; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Groin injuries, soccer, athletes, pain, muscle strength
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preventive treatment group (Experimental)
  Interventions: Other: preventive treatment group
- control group (No Intervention)

INTERVENTIONS:
Other: preventive treatment group — each athlete belonging to the preventive treatment group performed the protocol of preventive treatment 2 times a week, before or after the training session for five months
  Arms: preventive treatment group

SUMMARY:
Groin pain represents a common issue in football. Currently, there are no prevention protocols demonstrating real effectiveness. We aimed to investigate the possible positive effect of a prevention program for groin pain.Forty-two élite male athletes belonging to a youth academy of a professional football club were recruited in this prospective, randomized, controlled, single-blind, study.

ELIGIBILITY:
Inclusion Criteria:

* subjects between the ages of sixteen and eighteen, belonging to the youth sector of a professional club.

Exclusion Criteria:

* Presence of pain or injuries at the level of the hip-hip region at the initial assessment.

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Strength in the adductors | One day before the start of the physical protocol and one day after the end of the physical protocol
  The strength was evaluated in Newton during maximal voluntary isometric contraction used a dynamometer (Activforce 2)

SECONDARY OUTCOMES:
Pain in the hip joint | One day before the start of the physical protocol and one day after the end of the physical protocol
  The pain was rated using the Numeric Pain Rating Scale (NPRS) (0-10; 0 represents no pain and 10 represents maximum pain) during maximal voluntary isometric contraction (Copenhagen five-second squeeze test).
Groin pain | One day before the start of the physical protocol and one day after the end of the physical protocol
  The pain was rated using the Numeric Pain Rating Scale (NPRS) (0-10; 0 represents no pain and 10 represents maximum pain) during maximal voluntary isometric contraction (Copenhagen five-second squeeze test).
Range of motion (ROM) of the hip joint | One day before the start of the physical protocol and one day after the end of the physical protocol
  ROM was assessed using the distance (cm) from the head of the fibula to the edge of the bed (Bent Knee Fall Out Test)

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Genova, Genova, Italy

IPD SHARING:
Plan to Share IPD: No